CLINICAL TRIAL: NCT05873413
Title: RCT of a Combined MI Intervention to Address Bystander Behaviors in the Context of Alcohol Use
Brief Title: Motivations, Attitudes, and Perceptions Study
Acronym: MAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21912; R01AA029450 (NIH)
Record Dates: First submitted 2023-05-01; First posted 2023-05-24 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Drinking; Sexual Violence; Social Norms
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivate-the-Bystander (Active Comparator): A Zoom-based motivational interviewing prevention program that enhances knowledge, motivation, and skills for increased bystander behaviors.
  Interventions: Behavioral: Motivate-the-Bystander
- Motivate-the-Bystander+Alcohol (Experimental): A Zoom-based motivational interviewing prevention program that enhances knowledge, motivation, and skills for reduced alcohol use and increased bystander behaviors.
  Interventions: Behavioral: Motivate-the-Bystander+Alcohol
- Attention-only control (Placebo Comparator): A Zoom-based stress reduction program in which progressive muscle relaxation and other techniques are introduced and practiced.
  Interventions: Behavioral: Attention-only Control

INTERVENTIONS:
Behavioral: Motivate-the-Bystander — A Zoom-based motivational interviewing prevention program that enhances knowledge, motivation, and skills for increased bystander behaviors.
  Other Names: MTB
  Arms: Motivate-the-Bystander
Behavioral: Motivate-the-Bystander+Alcohol — A Zoom-based motivational interviewing prevention program that enhances knowledge, motivation, and skills for reduced alcohol use and increased bystander behaviors.
  Other Names: MTB+ALC
  Arms: Motivate-the-Bystander+Alcohol
Behavioral: Attention-only Control — A Zoom-based stress reduction program in which progressive muscle relaxation and other techniques are introduced and practiced.
  Other Names: Control
  Arms: Attention-only control

SUMMARY:
The goal of this clinical trial is to compare the impact of providing participants with

1. A recently developed protocol for motivating bystanders to intervene to help others who are in sexual risk situations (Motivate-the-Bystander) alone
2. Motivate-the-Bystander with an alcohol component focused on reducing drinking behaviors (Motivate-the-Bystander+Alcohol)
3. A control condition focused on reducing stress

The main questions it aims to answer are:

* Is Motivate-the-Bystander more effective than the attention control for increasing bystander behaviors?
* Is Motivate-the-Bystander+Alcohol more effective than MTB alone for increasing bystander behaviors?
* Is Motivate-the-Bystander+Alcohol more effective than Motivate-the-Bystander alone for decreasing alcohol use during bystander intervention opportunities?

Participants will:

* Complete online measures (e.g., self-reported bystander behaviors, past bystander training, history of bystander intervention attempts, sexual experiences, drinking behaviors, and other substance use behaviors)
* Complete either MTB, MTB+ALC, or the attention control condition online
* Complete the virtual reality simulation in the lab
* Complete electronic daily diary follow-up surveys about alcohol use and bystander intervention

DETAILED DESCRIPTION:
During young adulthood, an estimated one in five women experience sexual assault. The investigators seek to reduce this violence by motivating young adults to intervene with their peers to prevent sexual assault-an approach known as bystander intervention. Current bystander training is conducted in group sessions involving education about how to recognize and intervene in response to sexual risk situations. Although successful in changing knowledge and attitudes about sexual assault prevention, evaluations of these programs have rarely focused on changing actual bystander behaviors. Further, while bystander alcohol use is common in sexual risk situations, and undermines intervention attempts, alcohol consumption by bystanders is not explicitly targeted in existing intervention training programs. To address these gaps, the investigators will conduct a RCT comparing the efficacy of: 1) the recently developed bystander intervention, Motivate-the-Bystander (MTB), 2) MTB with an MI alcohol component (MTB+ALC), and 3) an attention control condition for reducing alcohol use and increasing bystander behaviors in response to sexual risk. Bystander behaviors will be assessed observationally during a virtual reality-based house party at 2 months post intervention. Participants' bystander behaviors, alcohol use, and relevant contextual variables will be assessed with an EMA measurement design using electronic daily diaries at baseline and weekly post intervention until month 9. The investigators expect that, compared to MTB alone and the control condition, MTB+ALC will produce significantly greater reductions in overall drinking and increases in prosocial bystander behaviors in a diverse sample of 450 young adults who are heavy drinkers. If the hypotheses are confirmed, results will support use of the combined MI-based bystander-alcohol intervention as an effective means of reducing drinking and motivating bystander behaviors among those at highest risk for sexual violence.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ages 18-25
* Heavy drinkers (as defined by using the AUDIT)
* English fluency
* Community members from Lancaster and surrounding counties in Nebraska
* Signed and dated consent form
* Stated willingness to comply with study procedures

Exclusion Criteria: This project does not have any pre-determined exclusion criteria beyond the need to meet inclusion criteria for the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol use | months 0-9
  Alcohol use quantity is assessed with electronic daily diaries weekly for 9 months.
Daily self-reports of bystander behavior | months 0-9
  Bystander behavior is assessed with electronic daily diaries weekly for 9 months.
Observational bystander behavior | 1-week follow-up
  Bystander behavior is assessed with a virtual environment called Bystander in Sexual Assault Virtual Environments (B-SAVE). Participants experience a virtual "house party" and are exposed to 10 situations in which they can intervene or not. Responses are recorded and coded for the presence and effectiveness of intervention attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Gervais, PhD, Principal Investigator — University of Nebraska Lincoln; David DiLillo, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska-Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers after the completion of the primary endpoint by contacting PIs DiLillo and Gervais or NIAAADA. Considerations for ensuring confidentiality of these shared data are described in Section 10.1.3. In addition, this study will comply with NIAAA Data Sharing Plans. All deidentified data will be shared with NIAAA for inclusion into the NIAAA Data Archive following the template provided by NIAAA.

DOCUMENTS (2):
  • Study Protocol (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT05873413/Prot_003.pdf
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT05873413/SAP_001.pdf